CLINICAL TRIAL: NCT04650737
Title: Single-Shot With Dexmedetomidine Versus Continuous Ultrasound-guided Erector Spinae Plane Block for Postoperative Pain Control After Percutaneous Nephrolithotomy Prospective Randomized Clinical Trial
Brief Title: Single-Shot With Dexmedetomidine Versus Continuous Ultrasound-guided Erector Spinae Plane Block for Postoperative Pain Control After Percutaneous Nephrolithotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ESPB in nephrolithotomy
Record Dates: First submitted 2020-11-13; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Both groups will receive Ultrasound guided ESPB before induction of general anesthesia
  * Single shot group (A):(20 patients) Patients in this group will receive 30 ml bupivacaine 0.25% plus 1ml of 1µg/kg Dexmedetomidine.
  * Continous infusion group (B):(20 patients) Patients in this group will receive 30 ml bupivacaine 0.25%plus 1ml normal salinefollowed by continuous infusion of 8ml / hour of 0.125% bupivacaine for 24 hrs
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (single shot,n=20) (Active Comparator): Patients in this group will receive 30 ml bupivacaine 0.25% plus 1ml of 1µg/kg Dexmedetomidine ;ultrasound guided ESPB
  Interventions: Drug: single shot ESBP with dexmedtomidine
- Group B (continous infusion,n=20) (Active Comparator): Patients in this group will receive 30 ml bupivacaine 0.25%plus 1ml normal salinefollowed by continuous infusion of 8ml / hour of 0.125% bupivacaine for 24 hrs;ESPB
  Interventions: Drug: continous ESPB

INTERVENTIONS:
Drug: single shot ESBP with dexmedtomidine — Patients in this group will receive errector spine plane block with 30 ml bupivacaine 0.25% plus 1ml of 1µg/kg Dexmedetomidine
  Arms: Group A (single shot,n=20)
Drug: continous ESPB — Patients in this group will receive erector spine plane block with 30 ml bupivacaine 0.25%plus 1ml normal salinefollowed by continuous infusion of 8ml / hour of 0.125% bupivacaine for 24 hrs.
  Arms: Group B (continous infusion,n=20)

SUMMARY:
The current study is designed to assess the efficacy of a single shot ESPB with Dexmedetomidineversus continuous ESPB in perioperative analgesia for PCNL. Both techniques are conducted for patients undergoing PCNL under GA.

DETAILED DESCRIPTION:
Successful perioperative pain management is one of the main goals of the whole anesthetic practice. Kidney Surgeries, especially those involving the renal pelvis warrant special analgesic considerations. This is due to the sensitivity of the renal pelvis to pain. Its sub-diaphragmatic position affects deep breathing and coughing. Which renders adequate analgesia an important factor for maintaining good respiratory force and depth postoperative and reduces respiratory complications like atelectasis.

The Use of a single mode of analgesia in these settings , like the use of parenteral opioids for example, provides significantly less analgesic effect and more complications including respiratory depression , PONV (postoperative nausea and vomiting ) , constipation , urine retention …etc.

The use of regional techniques as a part of multimodal pain management in these procedures provides superior analgesia and less complication rates.

This is added to high expectations of an easier perioperative course of PCNL (percutaneous nephrolithotomy) being and endoscopic procedure that does not involve a big skin incision. These expectations also include a short hospital stay. However PCNL is usually associated with significant pain and discomfort postoperatively. Various studies have been studying effects of integrating local and regional techniques in the perioperative pain management.

For Regional and local procedures of analgesia; Studies of Single Shot technique and catheter techniques has long been ongoing for many regional techniques for example like Pravertebral block and adductor canal block . These studies are conducted to determine the efficacy and adversities each technique.

Alpha-2 adrenoceptor agonists such as clonidine have been shown to increase the duration of peripheral nerve block . Dexmedetomidine is a more potent and selective α-2-adrenoceptor compared to clonidine . Peri-neural dexmedetomidine was evaluated in animal studies where it prolonged the duration of sensory and motor blocks of local anesthetics without any evidence of neurotoxicity for up to 14 days after initial administration . The use of perineuraldexmedetomidine prolong the duration of of sensory block, provide effective acute pain control after surgery and reduce the need for rescue analgesia in several nerve blocks like upper limb extremity blocks,Paravertebral block), tranversus abdominis plane (TAP) block and Erector spinae plane block.

Erector spinae plane block (ESPB) is a relatively novel procedure. The limited number of studies available show promising results as regards the efficacy of pain management in trunk surgeries and renal interventions. However the studies that clarify the different applications of ESPB, including the efficacy of a single shot versus a continuous block with an indwelling catheter, are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of age (18-50), ASA physical status I or II undergoing unilateral percutaneous nephrolithotomy

Exclusion Criteria:

* - Body mass index greater than 35 kg/m2.
* Pregnancy.
* Unstable coronary artery disease, congestive heart failure, or arrhythmias.
* Baseline heart rate (HR) less than 60 beats/min or baseline systolic blood pressure less than 100 mmHg.
* Pre-existing neurological deficits or neuropathy.
* Significant psychiatric or cognitive conditions interfering with consent or assessment.
* Significant renal impairment (creatinine above 2 mg/dl)
* Severe bronchopulmonary disease, including chronic obstructive pulmonary disease and obstructive sleep apnea.
* Known contraindications to peripheral nerve block, including local skin infections, bleeding diathesis, and coagulopathy.
* Allergies to local anesthetics, dexmedetomidine, or any component of multimodal analgesia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative Analgesia: | post-operative period(24 hours)
  "the time interval between extubation and the first request to postoperative analgesia

SECONDARY OUTCOMES:
Duration of sensory block | 24 hours
  the time interval between the onset of successful sensory block and the first request to postoperative analgesia
Visual analogue scale from 1 to 10,while 10 is the worst pain at rest and movement | 24 hours
  visual analogue scale during rest and movement

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Arshad Z, Zaidi SZ, Jamshaid A, Qureshi AH. Post operative pain control in percutaneous nephrolithotomy. J Pak Med Assoc. 2018 May;68(5):702-704. PMID 29885165
- [Background] Schug SA, Fry RA. Continuous regional analgesia in comparison with intravenous opioid administration for routine postoperative pain control. Anaesthesia. 1994 Jun;49(6):528-32. doi: 10.1111/j.1365-2044.1994.tb03528.x. PMID 8017600
- [Background] Choi SW, Cho SJ, Moon HW, Lee KW, Lee SH, Hong SH, Choi YS, Bae WJ, Ha US, Hong SH, Lee JY, Kim SW, Cho HJ. Effect of Intercostal Nerve Block and Nephrostomy Tract Infiltration With Ropivacaine on Postoperative Pain Control After Tubeless Percutaneous Nephrolithotomy: A Prospective, Randomized, and Case-controlled Trial. Urology. 2018 Apr;114:49-55. doi: 10.1016/j.urology.2017.12.004. Epub 2017 Dec 27. PMID 29288788
- [Background] Popping DM, Elia N, Marret E, Wenk M, Tramer MR. Clonidine as an adjuvant to local anesthetics for peripheral nerve and plexus blocks: a meta-analysis of randomized trials. Anesthesiology. 2009 Aug;111(2):406-15. doi: 10.1097/ALN.0b013e3181aae897. PMID 19602964
- [Background] Farag E, Argalious M, Abd-Elsayed A, Ebrahim Z, Doyle DJ. The use of dexmedetomidine in anesthesia and intensive care: a review. Curr Pharm Des. 2012;18(38):6257-65. doi: 10.2174/138161212803832272. PMID 22762468